CLINICAL TRIAL: NCT00063674
Title: Type 2 Diabetes Primary Prevention for At Risk Girls
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: T2DPPG (completed)
Record Dates: First submitted 2003-07-02; First posted 2003-07-03 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity; Diabetes Mellitus; Prediabetic State
Keywords: exercise; eating; dance; health education; obesity prevention; diabetes prevention; children
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Prediabetic State; Motor Activity; Health Education | interventions — Nutrition Assessment

INTERVENTIONS:
Behavioral: Nutrition Education
Behavioral: After-school dance class

SUMMARY:
Purpose: To evaluate two approaches to prevent obesity and type 2 diabetes in young girls.

The Need: We are experiencing an epidemic of childhood obesity. Rates of obesity have doubled to tripled in the past two decades, with the highest rates among poor and ethnic minority girls. Type 2 diabetes (what used to be called adult-onset diabetes) is now showing up in overweight children, and more children are manifesting precursors of heart disease and stroke.

Our Two Approaches:

1. A state-of-the-art nutrition education program with monthly newsletters mailed to girls and their parents and quarterly evening lectures/educational events at school sites, including cooking demonstrations and games to improve nutrition and increase physical activity.
2. After-school dance classes held five days per week all year long at school sites from the time school lets out until 6PM. Dance classes will include a 1-1.5 hour supervised homework study hall each day, and emphasize both traditional ethnic dances and popular dance.

Participants: Second, third and fourth grade girls and their families will be eligible to participate. All activities are free of charge. To be able to perform a valid evaluation, to be able to accommodate all girls at their own school, and to be fair about which girls receive which program, families who wish to participate will be randomly selected to participate in either one program or the other (nutrition education or dance classes). Each family will participate for two years.

Evaluation: Trained Stanford staff will perform all evaluation procedures with participating families in their own homes at the beginning and every six months. Families will be compensated for their participation.

ELIGIBILITY:
Second-, third- and fourth-grade girls, aged 7-10 years of age enrolled in one of the participating schools will be eligible. Our goal is to be as inclusive as possible. However, girls will not be eligible to participate if they:

* have been diagnosed with a chronic illness that affects their growth and/or weight (e.g., type 1 diabetes, hypothyroidism, inflammatory bowel disease)
* are taking medications potentially affecting their growth and/or weight (e.g., methylphenidate HCl, systemic steroids)
* have Asthma (not exclusionary alone) but have taken systemic steroids (oral, intravenous, or intramuscular) for a period of more than 21 days in the past year
* have a condition that limits their participation in physical activity enough that they are not able to participate in Physical Education at school (e.g., significant structural heart disease)
* are pregnant
* are unable to complete the informed consent process.

Ages: 7 Years to 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States